CLINICAL TRIAL: NCT05385120
Title: To Compare the Outcome of Temporary Portocaval Shunt During Recipient Hepatectomy Versus No Shunt in Adult Elective Live Donor Liver Transplantation- A Prospective Randomised Pilot Study
Brief Title: To Compare the Outcome of Temporary Portocaval Shunt During Recipient Hepatectomy Versus No Shunt in Adult Elective Live Donor Liver Transplantation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IEC/2021/91/MA04
Record Dates: First submitted 2022-03-29; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-03

CONDITIONS: Portosystemic Shunt
Keywords: Temporary Portocaval shunt; Recipient Hepatectomy; Liver transplantation

STUDY DESIGN:
Intervention Model Description: A Randomised Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A-Shunt group (Experimental): Patients who undergo temporary porto caval shunt (TPCS) during recipient hepatectomy in adult elective live donor liver transplantation
  Interventions: Procedure: Temporary Portocaval Shunt
- Group B-No Shunt group (No Intervention): Patients who donot undergo temporary porto caval shunt (TPCS) during recipient hepatectomy in adult elective live donor liver transplantation

INTERVENTIONS:
Procedure: Temporary Portocaval Shunt — In Temorary Portocaval Shunt Group (TPCS group), Hilar dissection( division of Hepatic artery, Bileduct) is followed by temporary portocaval shunt formation during recipient Hepatectomy.
  Arms: Group A-Shunt group

SUMMARY:
Temporary portocaval Shunt during recipient hepatectomy improves intra operative parameters and morbidity in LDLT recipients

DETAILED DESCRIPTION:
All patients satisfying the inclusion criteria, written informed consent will be taken and patients are randomized into intervention group ( Portocaval Shunt Group) and Non intervention group ( No Shunt Group).Patients from both the groups will be assessed for Hemodynamic parameters, Urine Output, Blood loss, blood products requirement , Duration of surgery during the procedure. They will be assessed for renal function, presence of sepsis, Morbidity, early graft dysfunction, ICU stay and total hospital stay in the post operative period.All patients will be followed up till discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

1) All Adult LDLT Recipients at ILBS, New Delhi

Exclusion Criteria:

1. Acute Liver Failure as an indication for transplant
2. Pediatric transplants
3. Presence of Yerdel grade III and grade IV Portal vein thrombosis
4. Presence of significant portosystemic shunting (greater than 10mm) in pre operative period.
5. Patients who have undergone TIPS procedure.
6. Hypercoagulable states like Budd-Chiari syndrome
7. Refusal to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-25 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure between two groups at fixed time points | T0- At the beginning of the procedure
  Systolic Blood pressure, Diastolic Blood Pressure and Mean Blood Pressure is measured in mmHg
Ionotropes requirement between two groups at fixed time points | T0- At the beginning of the procedure
  Noradrenaline and Vasopressin requirement in milliliter/hour
Lactate level between two groups at fixed time points | T0- At the beginning of the procedure
  Lactate levels are documented from Arterial Blood Gas analysis
Blood Pressure between two groups at fixed time points | T1- During procedure- Before portocaval shunt formation
  Systolic Blood pressure, Diastolic Blood Pressure and Mean Blood Pressure is measured in mmHg
Ionotropes requirement between two groups at fixed time points | T1- During procedure- Before portocaval shunt formation
  Noradrenaline and Vasopressin requirement in milliliter/hour
Lactate level between two groups at fixed time points | T1- During procedure- Before portocaval shunt formation
  Lactate levels are documented from Arterial Blood Gas analysis
Blood Pressure between two groups at fixed time points | T2- During procedure- Just Before Reperfusion of graft liver
  Systolic Blood pressure, Diastolic Blood Pressure and Mean Blood Pressure is measured in mmhg
Ionotropes requirement between two groups at fixed time points | T2- During procedure- Just Before Reperfusion of graft liver
  Noradrenaline and Vasopressin requirement in milliliter/hour
Lactate level between two groups at fixed time points | T2- During procedure- Just Before Reperfusion of graft liver
  Lactate levels are documented from Arterial Blood Gas analysis
Blood Pressure between two groups at fixed time points | T3- During procedure- 5 minutes after reperfusion of graft liver
  Systolic Blood pressure, Diastolic Blood Pressure and Mean Blood Pressure is measured in mmhg
Ionotropes requirement between two groups at fixed time points | T3- During procedure- 5 minutes after reperfusion of graft liver
  Noradrenaline and Vasopressin requirement in milliliter/hour
Lactate level between two groups at fixed time points | T3- During procedure- 5 minutes after reperfusion of graft liver
  Lactate levels are documented from Arterial Blood Gas analysis
Blood Pressure between two groups at fixed time points | T4- During procedure- Before closure of abdomen
  Systolic Blood pressure, Diastolic Blood Pressure and Mean Blood Pressure is measured in mmhg
Ionotropes requirement between two groups at fixed time points | T4- During procedure- Before closure of abdomen
  Noradrenaline and Vasopressin requirement in milliliter/hour
Lactate level between two groups at fixed time points | T4- During procedure- Before closure of abdomen
  Lactate levels are documented from Arterial Blood Gas analysis
Blood loss between two groups during intraoperative period | During Procedure
  Blood loss during the procedure is measured in milliliter
Duration of surgery between two groups. | During Procedure
  Duration between incision time to closure of abdomen is noted in minutes
Increase in creatinine levels of Increase 1.5-1.9 times from baseline in the post op period. | Number of days post transplantation procedure (upto 45 days)
  Serum Creatinine is measured in milligram per deciliter
≥0.3 mg/dl increase within 48 h or Urine output < 0.5 ml/kg/h for 6-12 h in the post op period. | Number of days post transplantation procedure (upto 45 days)
  Serum Creatinine is measured in milligram per deciliter
Urine output between two groups | During Transplantation procedure
  Urine output during the transplantation procedure is measured in milliliter

SECONDARY OUTCOMES:
To compare tolerance to enteral feed between two groups | Number of days post transplantation procedure (upto 45 days)
  Tolerance to NG feed is defined by absence of bloating, nausea, vomiting, abdominal distention or ileus
Endotoxin levels | Levels of Serum endotoxin levels in pre op and 12 hours after surgery
  Serum endotoxin levels increases in cases of bowel congestion and hemodynamic instability when portal vein is clamped during recipient hepatectomy
Number of patients with Early allograft dysfunction | For 5 consecutive days after day 7
  Early allograft dysfunction using criteria defined - total bilirubin >10 mg/dL, INR >1.6 and serum urea >100 mg/dL, for five consecutive days after day 7
Incidence of Morbidity | Number of days post transplantation procedure (upto 45 days)
  Morbidity is defined by Clavein Dindo Classification - >/=3. Sepsis as defined by Sepsis- 3 criteria, presence of 2 or more of the following 1.altered mentation, 2.respiratory rate ≥22 breaths/min 3.systolic blood pressure ≤100 mm Hg
Incidence of sepsis | Number of days post transplantation procedure (upto 45 days)
  Morbidity is defined by Clavein Dindo Classification - >/=3. Sepsis as defined by Sepsis- 3 criteria, presence of 2 or more of the following 1.altered mentation, 2.respiratory rate ≥22 breaths/min 3.systolic blood pressure ≤100 mm Hg
Number of days of ICU stay | Number of days post transplantation procedure (upto 45 days)
  Day patient shifted from ICU to ward is documented as total ICU stay. Day patient is discharged from hospital is documented for total hospital stay
Number of days of hospital stay | Number of days post transplantation procedure (upto 45 days)
  Day patient shifted from ICU to ward is documented as total ICU stay. Day patient is discharged from hospital is documented for total hospital stay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Figueras J, Llado L, Ramos E, Jaurrieta E, Rafecas A, Fabregat J, Torras J, Sabate A, Dalmau A. Temporary portocaval shunt during liver transplantation with vena cava preservation. Results of a prospective randomized study. Liver Transpl. 2001 Oct;7(10):904-11. doi: 10.1053/jlts.2001.27870. PMID 11679990
- [Result] Arzu GD, De Ruvo N, Montalti R, Masetti M, Begliomini B, Di Benedetto F, Rompianesi G, Di Sandro S, Smerieri N, D'Amico G, Vezzelli E, Iemmolo RM, Romano A, Ballarin R, Guerrini GP, De Blasiis MG, Spaggiari M, Gerunda GE. Temporary porto-caval shunt utility during orthotopic liver transplantation. Transplant Proc. 2008 Jul-Aug;40(6):1937-40. doi: 10.1016/j.transproceed.2008.06.001. PMID 18675094
- [Result] Ghinolfi D, Marti J, Rodriguez-Laiz G, Sturdevant M, Iyer K, Bassi D, Scher C, Schwartz M, Schiano T, Sogawa H, del Rio Martin J. The beneficial impact of temporary porto-caval shunt in orthotopic liver transplantation: a single center analysis. Transpl Int. 2011 Mar;24(3):243-50. doi: 10.1111/j.1432-2277.2010.01168.x. Epub 2010 Sep 28. PMID 20875093
- [Result] Kim JD, Choi DL. Beneficial impact of temporary portocaval shunt in living-donor liver transplantation with a difficult total hepatectomy. Transplant Proc. 2015 Apr;47(3):694-9. doi: 10.1016/j.transproceed.2014.12.036. PMID 25891713
- [Result] Pratschke S, Meimarakis G, Bruns CJ, Kaspar M, Prix N, Zachoval R, Guba M, Jauch KW, Loehe F, Angele MK. Temporary intraoperative porto-caval shunt: useless or beneficial in piggy back liver transplantation? Transpl Int. 2013 Jan;26(1):90-8. doi: 10.1111/tri.12007. Epub 2012 Nov 29. PMID 23237579